CLINICAL TRIAL: NCT00443456
Title: Long-Term Study For Amlodipine 10mg In Patients With Essential Hypertension For Whom Amlodipine 5mg Is Insufficiently Effective
Brief Title: Long Term Study Of Amlodipine 10mg With Hypertension For Whom Amlodipine 5mg Is Insufficient
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0531086
Record Dates: First submitted 2007-03-02; First posted 2007-03-06 (Estimated); Results first posted 2009-10-09 (Estimated); Last update posted 2009-10-28 (Estimated); Status verified 2009-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single (Experimental)
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Amlodipine — Two tablets of amlodipine 5 mg, Oral administration, Once daily for 44 weeks

SUMMARY:
To investigate the safety and efficacy of the long-term use of amlodipine 10 mg in subjects who will be able to enter a long-term study after completing the parent study "A double-blind comparative study between amlodipine 5 mg and 10 mg in patients with essential hypertension for whom amlodipine 5 mg is insufficiently effective" (Protocol No.: A0531085).

DETAILED DESCRIPTION:
NCT00415623 (protocol A0531085)

ELIGIBILITY:
Inclusion Criteria:

* Patients who had completed the preceding study A0531085, Phase III study, who the investigator judged to be able to further treatment of long term administration in terms of efficacy and safety
* Patients who had a treatment compliance rate of at least 80%

Exclusion Criteria:

* The patient who met the discontinuation criteria in the preceding study A0531085

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2007-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- Japan (9):
  - Pfizer Investigational Site, Chikushino-shi, Fukuoka
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Kitakyushu, Fukuoka
  - Pfizer Investigational Site, Yokohama, Kanagawa
  - Pfizer Investigational Site, Iruma, Saitama
  - Pfizer Investigational Site, Koshigaya, Saitama
  - Pfizer Investigational Site, Edogawa-ku, Tokyo
  - Pfizer Investigational Site, Setagaya-ku, Tokyo
  - Pfizer Investigational Site, Sumida-ku, Tokyo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0531086&StudyName=Long%20Term%20Study%20For%20Amlodipine%2010mg%20With%20Hypertension%20For%20Whom%20Amlodipine%205mg%20Is%20Insufficient

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Among subjects who had completed the preceding study (A0531085, NCT00415623), where either Amlodipine 5 mg or 10 mg was administered for 8 weeks, those who were considered to be eligible for enrollment in this long-term study, based on safety and efficacy of the preceding study and who had a treatment compliance rate of at least 80% were enrolled.
Groups:
- Amlodipine: All subjects who were treated with amlodipine at a dose of 10 mg during this long-term study.
Period: Overall Study
Arm/Group | Amlodipine
Started | 134
Completed | 116
Not Completed | 18
Not completed — Adverse Event | 16
Not completed — Move | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Amlodipine
Number analyzed (Participants) | 134
Age, Customized [Number; unit: participants]
  20 to 44 years | 13
  45 to 64 years | 65
  >=65 years | 56
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 73

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure From Baseline of the Preceding Study
Description: Value at each observation time point minus value at Week 0 (Week 0 was defined as baseline of the preceding study A0531085: NCT00415623.)
Time Frame: Week 0, 8 weeks, 10 weeks, 12 weeks, 16 weeks, 20 weeks, 24 weeks, 28 weeks, 32 weeks, 36 weeks, 40 weeks, 44 weeks, 48 weeks and 52 weeks
Population: Full Analysis Set, Last Observation Carried Forward
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Amlodipine: All subjects who were treated with amlodipine at a dose of 10 mg during this long-term study (A0531086: NCT00443456).
- The Preceding Study 5 mg Sub-set of This Long-term Study: Sub-set of subjects who received amlodipine 5 mg in the preceding study (A0531085: NCT00415623) then received 10 mg in this long-term study (A0531086: NCT00443456).
- The Preceding Study 10 mg Sub-set of This Long-term Study: Sub-set of subjects who received amlodipine 10 mg in the preceding study (A0531085: NCT00415623) then continued to receive 10 mg in this long-term study (A0531086: NCT00443456).
Arm/Group | Amlodipine | The Preceding Study 5 mg Sub-set of This Long-term Study | The Preceding Study 10 mg Sub-set of This Long-term Study
Number analyzed (Participants) | 134 | 69 | 65
mmHg
  Week 0: Baseline (Actual Value) | 148.8 (8.3) | 148.8 (8.0) | 148.8 (8.7)
  Week 8 | -8.7 (12.0) | -5.6 (12.9) | -12.0 (10.1)
  Week 10 | -14.8 (11.5) | -14.5 (11.3) | -15.0 (11.8)
  Week 12 | -15.6 (10.0) | -15.6 (9.7) | -15.7 (10.4)
  Week 16 | -16.7 (10.7) | -16.9 (10.5) | -16.4 (10.9)
  Week 20 | -15.8 (10.4) | -17.4 (11.1) | -14.1 (9.4)
  Week 24 | -15.4 (11.2) | -16.1 (10.5) | -14.6 (11.9)
  Week 28 | -14.7 (11.3) | -15.7 (11.7) | -13.6 (11.0)
  Week 32 | -13.8 (12.7) | -14.4 (12.4) | -13.2 (13.2)
  Week 36 | -13.4 (12.3) | -14.6 (12.0) | -12.2 (12.6)
  Week 40 | -13.9 (11.4) | -14.7 (11.6) | -13.0 (11.1)
  Week 44 | -15.7 (12.1) | -15.6 (12.5) | -15.8 (11.8)
  Week 48 | -15.3 (11.4) | -16.0 (11.6) | -14.5 (11.2)
  Week 52 | -15.6 (11.5) | -15.0 (11.7) | -16.3 (11.3)

2. Primary Outcome: Change in Systolic Blood Pressure From Baseline of This Long-term Study
Description: Value at each observation time point minus value at Week 8 (Week 8 was defined as baseline of this long-term study A0531086: NCT00443456.)
Time Frame: Week 8, 10 weeks, 12 weeks, 16 weeks, 20 weeks, 24 weeks, 28 weeks, 32 weeks, 36 weeks, 40 weeks, 44 weeks, 48 weeks and 52 weeks
Population: Full Analysis Set, Last Observation Carried Forward
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine | The Preceding Study 5 mg Sub-set of This Long-term Study | The Preceding Study 10 mg Sub-set of This Long-term Study
Number analyzed (Participants) | 134 | 69 | 65
mmHg
  Week 8: Baseline (Actual Value) | 140.1 (14.2) | 143.2 (15.7) | 136.8 (11.6)
  Week 10 | -6.0 (10.9) | -8.9 (11.2) | -3.0 (9.8)
  Week 12 | -6.9 (11.9) | -10.0 (13.6) | -3.7 (8.8)
  Week 16 | -8.0 (12.0) | -11.3 (13.3) | -4.4 (9.4)
  Week 20 | -7.1 (12.0) | -11.8 (12.7) | -2.1 (9.0)
  Week 24 | -6.7 (12.4) | -10.5 (12.7) | -2.6 (10.8)
  Week 28 | -6.0 (13.0) | -10.1 (13.9) | -1.6 (10.3)
  Week 32 | -5.1 (12.2) | -8.8 (13.0) | -1.2 (9.9)
  Week 36 | -4.7 (12.6) | -9.0 (13.2) | -0.2 (10.4)
  Week 40 | -5.2 (13.7) | -9.1 (14.9) | -1.0 (10.9)
  Week 44 | -7.0 (12.6) | -10.0 (14.1) | -3.8 (10.0)
  Week 48 | -6.6 (13.4) | -10.4 (14.4) | -2.5 (10.9)
  Week 52 | -6.9 (13.0) | -9.4 (14.0) | -4.3 (11.4)

3. Primary Outcome: Change in Diastolic Blood Pressure From Baseline of the Preceding Study
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Full Analysis Set, Last Observation Carried Forward
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine | The Preceding Study 5 mg Sub-set of This Long-term Study | The Preceding Study 10 mg Sub-set of This Long-term Study
Number analyzed (Participants) | 134 | 69 | 65
mmHg
  Week 0: Baseline (Actual Value) | 86.3 (10.2) | 87.6 (10.0) | 84.8 (10.2)
  Week 8 | -3.1 (8.8) | -1.8 (9.4) | -4.5 (7.9)
  Week 10 | -6.4 (7.9) | -6.6 (7.7) | -6.3 (8.1)
  Week 12 | -6.9 (7.6) | -7.7 (7.9) | -6.0 (7.2)
  Week 16 | -7.3 (8.0) | -8.4 (8.0) | -6.2 (7.9)
  Week 20 | -7.2 (8.0) | -7.9 (8.0) | -6.4 (7.9)
  Week 24 | -6.8 (8.1) | -7.1 (8.6) | -6.5 (7.6)
  Week 28 | -6.8 (8.3) | -7.8 (8.9) | -5.7 (7.5)
  Week 32 | -6.8 (8.6) | -7.1 (8.5) | -6.5 (8.8)
  Week 36 | -6.5 (8.4) | -7.4 (7.9) | -5.5 (8.9)
  Week 40 | -6.8 (8.7) | -7.2 (9.6) | -6.3 (7.8)
  Week 44 | -7.3 (8.0) | -7.6 (8.2) | -6.9 (7.8)
  Week 48 | -7.2 (8.8) | -7.3 (9.4) | -7.0 (8.2)
  Week 52 | -7.9 (8.5) | -8.2 (7.9) | -7.7 (9.2)

4. Primary Outcome: Change in Diastolic Blood Pressure From Baseline of This Long-term Study
Description: as for outcome 2
Time Frame: as for outcome 2
Population: Full Analysis Set, Last Observation Carried Forward
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine | The Preceding Study 5 mg Sub-set of This Long-term Study | The Preceding Study 10 mg Sub-set of This Long-term Study
Number analyzed (Participants) | 134 | 69 | 65
mmHg
  Week 8: Baseline (Actual Value) | 83.1 (11.5) | 85.8 (11.8) | 80.3 (10.5)
  Week 10 | -3.3 (7.2) | -4.8 (7.5) | -1.7 (6.6)
  Week 12 | -3.7 (7.3) | -5.8 (8.1) | -1.5 (5.6)
  Week 16 | -4.2 (7.9) | -6.5 (8.3) | -1.7 (6.6)
  Week 20 | -4.1 (7.5) | -6.1 (8.3) | -1.9 (5.8)
  Week 24 | -3.7 (8.4) | -5.3 (8.4) | -2.0 (8.2)
  Week 28 | -3.7 (8.3) | -6.0 (8.8) | -1.2 (6.9)
  Week 32 | -3.6 (8.4) | -5.2 (8.3) | -1.9 (8.3)
  Week 36 | -3.3 (9.2) | -5.6 (9.1) | -0.9 (8.7)
  Week 40 | -3.6 (9.1) | -5.4 (9.8) | -1.7 (8.0)
  Week 44 | -4.1 (8.3) | -5.8 (8.7) | -2.3 (7.4)
  Week 48 | -4.1 (8.7) | -5.5 (9.5) | -2.5 (7.6)
  Week 52 | -4.8 (9.6) | -6.3 (9.5) | -3.2 (9.5)

5. Other Pre Specified Outcome: Change in Systolic Blood Pressure From Baseline of the Preceding Study in Treatment Groups With or Without Concomitant Antihypertensive Agent
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Full Analysis Set, Observed Case, n=number of subjects with evaluable data in group with concomitant treatment, without concomitant treatment, respectively.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Subjects With Concomitant Antihypertensive Agent: Subjects receiving 10 mg amlodipine who were treated with concomitant antihypertensive agent at Week 12 or later.
- Subjects Without Concomitant Antihypertensive Agent: Subjects receiving 10 mg amlodipine who did not use concomitant antihypertensive agent during this long-term study (A0531086: NCT00443456).
Arm/Group | Subjects With Concomitant Antihypertensive Agent | Subjects Without Concomitant Antihypertensive Agent
Number analyzed (Participants) | 13 | 121
mmHg
  Week 0: Baseline (Actual Value) | 153.9 (10.8) | 148.3 (7.9)
  Week 8 (n=13, 121) | -4.8 (8.1) | -9.1 (12.3)
  Week 10 (n=13, 118) | -13.8 (8.7) | -14.8 (11.8)
  Week 12 (n=12, 119) | -13.5 (8.0) | -15.8 (9.9)
  Week 16 (n=12, 117) | -17.2 (8.9) | -16.4 (10.5)
  Week 20 (n=12, 116) | -10.8 (6.0) | -16.1 (10.3)
  Week 24 (n=11, 113) | -13.8 (14.0) | -14.8 (10.2)
  Week 28 (n=12, 111) | -15.1 (10.9) | -13.6 (10.4)
  Week 32 (n=12, 111) | -4.8 (13.9) | -14.0 (11.7)
  Week 36 (n=11, 108) | -4.8 (13.2) | -13.1 (11.5)
  Week 40 (n=12, 108) | -9.6 (8.3) | -13.6 (10.9)
  Week 44 (n=11, 108) | -13.7 (8.3) | -15.4 (12.0)
  Week 48 (n=9, 107) | -11.1 (12.5) | -15.3 (10.6)
  Week 52 (n=9, 106) | -10.8 (8.5) | -15.9 (11.0)

6. Other Pre Specified Outcome: Change in Systolic Blood Pressure From Baseline of This Long-term Study in Treatment Groups With or Without Concomitant Antihypertensive Agent
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Subjects With Concomitant Antihypertensive Agent | Subjects Without Concomitant Antihypertensive Agent
Number analyzed (Participants) | 13 | 121
mmHg
  Week 8: Baseline (Actual Value) | 149.1 (15.1) | 139.2 (13.8)
  Week 10 (n=13, 118) | -9.0 (9.0) | -5.9 (11.2)
  Week 12 (n=12, 119) | -8.4 (9.2) | -6.9 (12.2)
  Week 16 (n=12, 117) | -12.0 (9.8) | -7.6 (12.3)
  Week 20 (n=12, 116) | -5.6 (8.6) | -7.3 (12.3)
  Week 24 (n=11, 113) | -9.2 (15.4) | -6.2 (12.1)
  Week 28 (n=12, 111) | -9.9 (13.1) | -5.0 (12.7)
  Week 32 (n=12, 111) | 0.4 (17.5) | -5.3 (11.5)
  Week 36 (n=11, 108) | 0.2 (18.7) | -4.5 (12.0)
  Week 40 (n=12, 108) | -4.5 (11.2) | -5.2 (14.1)
  Week 44 (n=11, 108) | -9.1 (13.2) | -7.1 (12.6)
  Week 48 (n=9, 107) | -7.3 (17.4) | -7.0 (13.2)
  Week 52 (n=9, 106) | -7.1 (13.9) | -7.5 (13.1)

7. Other Pre Specified Outcome: Change in Diastolic Blood Pressure From Baseline of the Preceding Study in Treatment Groups With or Without Concomitant Antihypertensive Agent
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Subjects With Concomitant Antihypertensive Agent | Subjects Without Concomitant Antihypertensive Agent
Number analyzed (Participants) | 13 | 121
mmHg
  Week 0: Baseline (Actual Value) | 85.9 (12.4) | 86.3 (10.0)
  Week 8 (n=13, 121) | 0.3 (9.9) | -3.5 (8.6)
  Week 10 (n=13, 118) | -3.6 (9.1) | -6.6 (7.7)
  Week 12 (n=12, 119) | -4.8 (9.7) | -7.0 (7.4)
  Week 16 (n=12, 117) | -4.9 (9.2) | -7.6 (8.0)
  Week 20 (n=12, 116) | -2.5 (9.3) | -7.7 (7.9)
  Week 24 (n=11, 113) | -2.9 (10.3) | -6.9 (8.1)
  Week 28 (n=12, 111) | -3.2 (7.5) | -6.9 (8.6)
  Week 32 (n=12, 111) | 1.7 (7.6) | -7.4 (8.6)
  Week 36 (n=11, 108) | 2.1 (8.6) | -7.0 (8.2)
  Week 40 (n=12, 108) | 0.8 (6.8) | -7.3 (8.8)
  Week 44 (n=11, 108) | -2.4 (7.0) | -7.5 (8.2)
  Week 48 (n=9, 107) | -0.8 (9.4) | -7.5 (9.0)
  Week 52 (n=9, 106) | -2.7 (7.3) | -8.4 (8.9)

8. Other Pre Specified Outcome: Change in Diastolic Blood Pressure From Baseline of This Long-term Study in Treatment Groups With or Without Concomitant Antihypertensive Agent
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Subjects With Concomitant Antihypertensive Agent | Subjects Without Concomitant Antihypertensive Agent
Number analyzed (Participants) | 13 | 121
mmHg
  Week 8: Baseline (Actual Value) | 86.2 (11.8) | 82.8 (11.4)
  Week 10 (n=13, 118) | -3.9 (5.4) | -3.3 (7.5)
  Week 12 (n=12, 119) | -5.0 (4.9) | -3.7 (7.6)
  Week 16 (n=12, 117) | -5.1 (5.0) | -4.2 (8.2)
  Week 20 (n=12, 116) | -2.8 (6.4) | -4.4 (7.7)
  Week 24 (n=11, 113) | -4.0 (8.4) | -3.6 (8.7)
  Week 28 (n=12, 111) | -3.5 (8.6) | -3.6 (8.4)
  Week 32 (n=12, 111) | 1.5 (9.8) | -4.2 (8.4)
  Week 36 (n=11, 108) | 2.3 (11.8) | -3.8 (9.2)
  Week 40 (n=12, 108) | 0.6 (6.6) | -4.1 (9.6)
  Week 44 (n=11, 108) | -3.4 (9.2) | -4.4 (8.5)
  Week 48 (n=9, 107) | -1.9 (11.0) | -4.6 (8.9)
  Week 52 (n=9, 106) | -3.8 (10.2) | -5.4 (10.1)

9. Primary Outcome: Number of Subjects Whose Blood Pressure Reached Target Blood Pressure Reduction Value
Description: Target blood pressure reduction value in accordance with Japanese Society of Hypertension Guidelines for the Management of Hypertension 2004: For <= 64 years old: systolic blood pressure below 130 mmHg and diastolic blood pressure below 85 mmHg; For >= 65 years old: systolic blood pressure below 140 mmHg and diastolic blood pressure below 90 mmHg
Time Frame: 8 weeks, 10 weeks, 12 weeks, 16 weeks, 20 weeks, 24 weeks, 28 weeks, 32 weeks, 36 weeks, 40 weeks, 44 weeks, 48 weeks and 52 weeks
Population: Full Analysis Set, Last Observation Carried Forward
Measure: Number; unit: participants
Arm/Group | Amlodipine | The Preceding Study 5 mg Sub-set of This Long-term Study | The Preceding Study 10 mg Sub-set of This Long-term Study
Number analyzed (Participants) | 134 | 69 | 65
participants
  Week 8 | 41 | 15 | 26
  Week 10 | 59 | 27 | 32
  Week 12 | 64 | 30 | 34
  Week 16 | 62 | 29 | 33
  Week 20 | 65 | 35 | 30
  Week 24 | 64 | 32 | 32
  Week 28 | 54 | 30 | 24
  Week 32 | 53 | 23 | 30
  Week 36 | 56 | 32 | 24
  Week 40 | 56 | 29 | 27
  Week 44 | 58 | 26 | 32
  Week 48 | 58 | 31 | 27
  Week 52 | 63 | 29 | 34

10. Primary Outcome: Number of Subjects Whose Blood Pressure Reached Target Blood Pressure Reduction Value and Systolic Blood Pressure Had Decreased by 10 mmHg or More From Baseline in the Preceding Study
Description: as for outcome 9
Time Frame: as for outcome 9
Population: Full Analysis Set, Last Observation Carried Forward
Measure: Number; unit: participants
Arm/Group | Amlodipine | The Preceding Study 5 mg Sub-set of This Long-term Study | The Preceding Study 10 mg Sub-set of This Long-term Study
Number analyzed (Participants) | 134 | 69 | 65
participants
  Week 8 | 36 | 13 | 23
  Week 10 | 55 | 25 | 30
  Week 12 | 60 | 29 | 31
  Week 16 | 59 | 28 | 31
  Week 20 | 62 | 35 | 27
  Week 24 | 60 | 30 | 30
  Week 28 | 54 | 30 | 24
  Week 32 | 50 | 22 | 28
  Week 36 | 54 | 32 | 22
  Week 40 | 52 | 27 | 25
  Week 44 | 57 | 25 | 32
  Week 48 | 56 | 30 | 26
  Week 52 | 60 | 28 | 32

11. Other Pre Specified Outcome: Number of Subjects Whose Blood Pressure Reached Target Blood Pressure Reduction Value in Treatment Groups With or Without Concomitant Antihypertensive Agent
Description: as for outcome 9
Time Frame: as for outcome 9
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Subjects With Concomitant Antihypertensive Agent | Subjects Without Concomitant Antihypertensive Agent
Number analyzed (Participants) | 13 | 121
participants
  Week 8 (n=13, 121) | 2 | 39
  Week 10 (n=13, 118) | 3 | 54
  Week 12 (n=12, 119) | 4 | 59
  Week 16 (n=12, 117) | 4 | 56
  Week 20 (n=12, 116) | 3 | 59
  Week 24 (n=11, 113) | 2 | 57
  Week 28 (n=12, 111) | 2 | 46
  Week 32 (n=12, 111) | 2 | 46
  Week 36 (n=11, 108) | 2 | 45
  Week 40 (n=12, 108) | 1 | 48
  Week 44 (n=11, 108) | 1 | 49
  Week 48 (n=9, 107) | 1 | 49
  Week 52 (n=9, 106) | 1 | 54

12. Other Pre Specified Outcome: Number of Subjects Whose Blood Pressure Reached Target Blood Pressure Reduction Value and Systolic Blood Pressure Had Decreased by 10 mmHg or More From Baseline in the Preceding Study in Treatment Groups With or Without Concomitant Antihypertensive Agent
Description: as for outcome 9
Time Frame: as for outcome 9
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Subjects With Concomitant Antihypertensive Agent | Subjects Without Concomitant Antihypertensive Agent
Number analyzed (Participants) | 13 | 121
participants
  Week 8 (n=13, 121) | 1 | 35
  Week 10 (n=13, 118) | 3 | 50
  Week 12 (n=12, 119) | 4 | 55
  Week 16 (n=12, 117) | 4 | 53
  Week 20 (n=12, 116) | 3 | 56
  Week 24 (n=11, 113) | 2 | 53
  Week 28 (n=12, 111) | 2 | 46
  Week 32 (n=12, 111) | 2 | 43
  Week 36 (n=11, 108) | 2 | 43
  Week 40 (n=12, 108) | 1 | 44
  Week 44 (n=11, 108) | 1 | 48
  Week 48 (n=9, 107) | 1 | 47
  Week 52 (n=9, 106) | 1 | 51

ADVERSE EVENTS:
Arm/Group | Amlodipine
Serious Adverse Events (participants affected / at risk) | 8/134
Other Adverse Events (participants affected / at risk) | 50/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amlodipine (N=134)
Angina unstable (Cardiac disorders) | 1
Atrioventricular block (Cardiac disorders) | 1
Sick sinus syndrome (Cardiac disorders) | 1
Fall (Injury, poisoning and procedural complications) | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gum neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral infarction (Nervous system disorders) | 1
Dizziness postural (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Amlodipine (N=134)
Oedema peripheral (General disorders) | 15
Nasopharyngitis (Infections and infestations) | 33
Back pain (Musculoskeletal and connective tissue disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.